CLINICAL TRIAL: NCT06373445
Title: Therapeutic Effect of Repetitive Transcranial Magnetic Stimulation on Sleep Disorders in Fibromyalgia Patients : A Double Blinded, Randomized Clinical Trial
Brief Title: Interventional Neuromodulation in Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Marwa Y Badr, MD, Principal investigator, Tanta University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 36264PR596
Record Dates: First submitted 2024-04-09; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Neuromodulation and Sleep Disorders
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: participants randomly allocated to either no, one, some or all interventions simultaneously
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): The transcranial magnetic stimulation sessions were carried out using the MAGSTIM TMS equipment (Company Limited, Whitland, wales, UK). The investigators used the figure of eight or butterfly coil. The experimental group received real rTMS as follow: The intensity of the stimulus employed in treatment has used the motor threshold (MT) as the basic measure. The MT is used as a measurement index because the motor cortex is the only brain region which gives an easily detected signal [muscle twitch] when depolarized.The main stimulation parameters were 24 trains at120% of motor threshold for 60 seconds at 1 Hz and a 45-second interval between trains. The investigators subsequently provided a total of 1,200 pulses at each of the 20 sessions. The stimulation area was the right dorsolateral prefrontal area that was defined as the region 5 cm rostral in the same sagittal plane as the optimal site for MT production in the first dorsal interosseous
  Interventions: Device: repetitive transcranial magnetic stimulation active stimulation
- control group (Sham Comparator): The control group received sham rTMS as in the experimental group; however, sham current was with the coil placed perpendicular to the with the coil placed perpendicular to the scalp. The investigator responsible for delivering rTMS had no contact with the patients, ensuring a double-blind procedure.
  Interventions: Device: repetitive transcranial magnetic stimulation sham stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation active stimulation — This study was conducted on 20 eligible fibromyalgia patients with sleep disorders. They were randomized to have 20 sessions of active rTMS (1 Hz, 120% of resting motor threshold with total 1200 pules /session) over the right dorsolateral prefrontal area (DLPFC) for 5 sessions/week for 4 weeks.
  Arms: Active group
Device: repetitive transcranial magnetic stimulation sham stimulation — This study was conducted on 20 eligible fibromyalgia patients with sleep disorders. They were randomized to have 20 sessions of sham rTMS (1 Hz, 120% of resting motor threshold with total 1200 pules /session) over the right dorsolateral prefrontal area (DLPFC) for 5 sessions/week for 4 weeks.
  Arms: control group

SUMMARY:
This study was conducted on 40 eligible fibromyalgia patients with sleep disorders. They were randomized to have 20 sessions of active or sham rTMS (1 Hz, 120% of resting motor threshold with total 1200 pules /session) over the right dorsolateral prefrontal area (DLPFC) for 5 sessions/week for 4 weeks. All participants were subjected to baseline evaluation with Fibromyalgia Impact Questionnaire, polysomnography, sleep quality and sleep characteristics assessment using the Pittsburgh Sleep Quality Index and The Medical Outcomes Study Sleep Scale respectively.FM patients were reevaluated at 1, 3 months after the end of rTMS sessions.

DETAILED DESCRIPTION:
This is a prospective double randomized controlled trial that was conducted in Tanta and Assiut University hospitals during the period from 1st October 2022 to the end of March 2023. Sixty four 64 patients with fibromyalgia were recruited from outpatient clinics of Physical Medicine, Rheumatology and Rehabilitation and Neuropsychiatry Departments, Tanta and Assiut University Hospitals. The diagnosis of fibromyalgia was done according to American College of Rheumatology criteria or other standard criteria.

Twenty two cases didn't meet the inclusion and exclusion criteria were excluded: 8 of them had systemic diseases, 5 patients refuse to participate, 4 had contraindication for magnetic stimulation, and 5 cases had primary psychiatric disorders. Forty two cases were eligible and allocated into one of the two groups (1:1 ratio) active rTMS group and sham rTMS group. One case from each group didn't complete the follow up study due to headache and the remaining 20 cases in each group completed the study.

Each patient was subjected to history taking including age of symptoms onset and duration, complete clinical and neurological examination neurological examinations. Fibromyalgia Impact Questionnaire (FIQ) was assessed at base line. Besides, baseline Sleep quality and sleep characteristics assessment using the Pittsburgh Sleep Quality Index (PSQI) and The Medical Outcomes Study Sleep Scale (MOS Sleep Scale) respectively .

Randomization All qualified members were haphazardly doled out to one of the two groups. Assignment concealment was done utilizing serially numbered closed, enigmatic envelopes. Each patient was given a serial number from a computer-created randomization table and was put within the suitable group after opening the congruent closed envelope. Counseling for participation was conducted before enrollment.

Procedure of repetitive transcranial magnetic stimulation (rTMS):

Forty two fibromyalgia patients who had regular appropriate trial of medical treatment for at least 3 months, underwent 20 sessions of 30 minutes duration for each session of low frequency real or active rTMS at a rate of 5 sessions per week over 4 consecutive weeks, they were carried out by a qualified expert in this field. The transcranial magnetic stimulation sessions were carried out using the MAGSTIM TMS equipment (Company Limited, Whitland, wales, UK). The apparatus consists of a stimulator and a coil connected to the stimulator by a thick , insulated cable. The investigators used the figure of eight or butterfly coil. It's constructed of two circular coils, about 7 cm in diameter, mounted next to each other.

The experimental group received real rTMS as follow: The intensity of the stimulus employed in treatment has used the motor threshold (MT) as the basic measure. To determine the MT, the coil is placed over the motor cortex and moved until the smallest possible impulse produces a visible movement of the thumb, wrist or fingers. The MT is used as a measurement index because the motor cortex is the only brain region which gives an easily detected signal [muscle twitch] when depolarized . The main stimulation parameters were 24 trains at120% of motor threshold for 60 seconds at 1 Hz and a 45-second interval between trains. The investigators subsequently provided a total of 1,200 pulses at each of the 20 sessions. The stimulation area was the right dorsolateral prefrontal area that was defined as the region 5 cm rostral in the same sagittal plane as the optimal site for MT production in the first dorsal interosseous .

The sham rTMS group received the same protocol of active group however the coil held perpendicular to the scalp. The investigator responsible for delivering rTMS had no contact with the patients, ensuring a double-blind procedure.

Polysomnography Evaluation:

All patients at baseline on medical ttt alone(before rTMS sessions), were subjected to one night Polysomnography:. PSG was performed by a Nihon Kohden corporation (1-31-4 Nishiochiai, Shinjuku-Ku, Tokyo 161-8560,Japan, SN: 04142: 2018). The PSG involved EEG channels montages (O1/A2, C3/A2, C4/A1 and O2/A1), electrooculography (LOC-A1/A2 and ROC-A1/A2), surface tibial and submental EMG(electromyography), and modified V2 lead ECG. Thermal airflow sensors (thermistors) were utilized for nasal and oral signals and the amplifier was connected for tracheal sound appraisal. Chest and abdominal endeavors were measured by double thoracoabdominal RIP (respiratory inductance plethysmography) belts. PSG parameters (Sleep latency, Apnea hypopnea index, Sleep efficiency , Arousal index , Total sleep time(TST), Wake after sleep onset, Wake % TST, N1 % TST, N2%TST, N3%TST, REM(rapid eye movement) %TST, PLMs(periodic limb movements) index) were scored by a PSG technician and interpreted by a trained, expert sleep medicine physician according to The American Academy of Sleep Medicine guidelines . Apneas and hypopneas were defined according to standard methods .

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 to 50 years.
* Regular appropriate trial of medical treatment for at least 3 months.
* Educated participants at least 12 years.

Exclusion Criteria:

* Inflammatory rheumatic disease, auto immune disease or other painful disorders.
* Any uncontrolled clinical disease (such as thyroid, cardiovascular, pulmonary, hematological or renal disease) that affect the cognition.
* pregnancy, lactation.
* Contra indications for transcranial magnetic stimulation-a history of seizures, brain trauma, brain surgery or intracranial hypertension, a pace maker or other metallic implants.
* Past history of major sleep disorders(narcolepsy, parasomnia or sleep apnea).
* Illicit drug or alcohol abuse.
* Inability to cooperate with the questionnaire survey.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | baseline and one month after the end of sessions
  Improvement of sleep quality in patients with fibromyalgia to treatment with repetitive transcranial magnetic stimulation sessions.
The Medical Outcomes Study Sleep Scale (MOS ) | baseline and one month after the end of sessions
  Improvement of sleep characteristics in patients with fibromyalgia to treatment with repetitive transcranial magnetic stimulation sessions.
polysomnography | baseline and one month after the end of sessions
  Improvement of objective sleep parameter abnormalities in patients with fibromyalgia to treatment with repetitive transcranial magnetic stimulation sessions.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | "through study completion, an average of 6 months after the end of sessions"
  stabilization of obvious improvement of sleep quality in patients with fibromyalgia after rTMS sessions with better quality of life
The Medical Outcomes Study Sleep Scale (MOS) | "through study completion, an average of 6 months after the end of sessions"
  stabilization of obvious improvement of sleep characteristics in patients with fibromyalgia after rTMS sessions with better quality of life
polysomnography | "through study completion, an average of 6 months after the end of sessions"
  stabilization of obvious improvement of objective sleep parameter abnormalities in patients with fibromyalgia after rTMS sessions with better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Eman Khedr, MD neurology, Study Director — Assiut University
Locations (1):
- Faculty of medicine, Tanta, ElGharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after deidentification (texts, tables, figures and appendices)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 6 months
Access Criteria: controlled data analysis, third party